CLINICAL TRIAL: NCT01186952
Title: Effects of an Exercise Program Combined or Not With Nutritional intErvention on Total Fat, Epicardial Fat and Metabolic Profile of Obese and Overweight Adults With tyPe 2 Diabetes (The PEP-2 Study)
Brief Title: Exercise Program Combined or Not With Nutritional intErvention in Adults With tyPe 2 Diabetes
Acronym: PEP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, MD, PhD, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RRL-01-2010
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Overweight; Obesity; Type 2 Diabetes
Keywords: overweight; obesity; type 2 diabetes; caloric restriction; exercise program; epicardial fat
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Optimized usual care (No Intervention): participants will attend one visit with the dietician (30mn) and the physical activity specialist (30mn) when they will be given Canadian guidelines pamphlets for physical activity and food consumption. They will also receive a phone call once a month to discuss about issues in guidelines following.
- Diet intervention alone (Active Comparator): Participants will attend one visit with the physical activity specialist (30mn) when they will receive the physical activity guidelines. Monthly phone call will be make to discuss about issues in physical activity guidelines following.These individuals will also be enrolled in a supervised caloric restriction program. They will have to visit the dietician once a week for the first months and then twice a month for 3 months. The diet intervention will focus on a low fat diet. At each session participants will be weighed and taken the blood pressure.
  Interventions: Behavioral: Caloric restriction
- diet intervention and exercise program (Active Comparator): Participants will attend diet intervention as described for group 2. They will also follow a supervised exercise program three days per week for 4 months. The exercise training is an interval high intensity aerobic (85-90% heart rate reserve) program with resistance exercises (15RM, 2-3 repetitions). Each session will last one hour. At the end of month 1, 2, and 3, all participants will receive the SWA armband for 7 days to record physical activity and estimate energy expenditure.
  At the end of Month 4, all participants will attend a study visit for repeat baseline testing.
  Interventions: Behavioral: Diet intervention and structured exercise training program

INTERVENTIONS:
Behavioral: Caloric restriction — The caloric restriction diet will follow the Canadian Diabetes Association guidelines and be nutritionally balanced with a reduced total fat as well as saturated content.
  Other Names: Structured diet intervention (caloric restriction)
  Arms: Diet intervention alone
Behavioral: Diet intervention and structured exercise training program — Participants will follow the diet intervention previously described and a supervised physical activity program. The supervised exercise training sessions will take place three times a week for 4 months. Each session will last 1hour and will include aerobic exercise and resistance training. The aerobic training program will be treadmills intervals exercise at 50-70 % of heart rate reserve(HRR) the first month and 85-90% of HRR from the second to the fourth month. The resistance training programme will consist of two to three sets of 12 repetitions of the following exercises: leg press, chest press, lat pulldown, shoulder press, biceps curl, triceps extension.
  Other Names: diet intervention and exercise program.
  Arms: diet intervention and exercise program

SUMMARY:
Inactivity and excess energy consumption are leading causes of obesity and type 2 diabetes which are associated with increased cardio-metabolic risk. In order to reduce the cardiovascular risk associated with type 2 diabetes, the Canadian Diabetes Association guidelines (2008) recommends weight loss through caloric restriction and structured physical activity. However, the comparative effects of different methods to obtain caloric deficit for weight loss remains to be elucidated. The main objective of this study is to assess the impact of two strategies of caloric deficit: diet alone or diet and exercise on total fat mass, epicardial fat and cardiovascular risk factors in overweight and obese adults with type 2 diabetes and at high risk of cardiovascular disease.

DETAILED DESCRIPTION:
Type 2 diabetes is mainly caused by excess body weight due to lack of physical activity and high amount of calories consumption. Individuals with type 2 diabetes demonstrated increased risk of cardiovascular disease compared to non diabetic. Studies showed a cardiovascular risk reduction after weight loss among individuals at risk through lifestyle modification: increase physical activity and low calorie diet.

Favourable effects of weight loss on cardiovascular risk are mainly due to total body fat reduction. However, the location of body fat excess has also some important implications. It is now well known that abdominal (visceral) and ectopic fat accumulation (e.g. hepatic fat, epicardial fat, etc.) are more related to an unfavorable cardio-metabolic profile than total fat mass. It has been demonstrated that a moderate weight loss obtained with physical activity or caloric restriction is related to a significant reduction of ectopic fat mass. However, ectopic fat measurement remains problematic due to lack of standardization and safety issues (X-ray). Epicardial fat thickness measured by simple echocardiography is a reliable method to evaluate ectopic fat accumulation.

Little research have been done to assess the effect of different methods of weight loss on total fat as well as ectopic fat specifically epicardial adipose tissue among individuals with type 2 diabetes. The objective of this study is to compare to a control group with detailed advice the impact of two structured strategies of caloric deficit: diet alone or diet and exercise on total fat mass, epicardial fat and cardiovascular risk factors in overweight and obese adults with type 2 diabetes and at high risk of cardiovascular disease.

The participants to the present study will be free-living adults overweight and obese with type 2 diabetes and at high risk of cardiovascular disease as determined by a Framingham risk score above 15% or the presence of two or more cardiovascular risk factors.

Participants will attend a screening study visit to confirm eligibility criteria (anthropometric variables, blood pressure, complete physical examination, coronary heart disease diagnostic by echocardiogram, physical activity aptitude).

After enrollment, a baseline visit will consist in series of data collection such as : anthropometric variables, blood pressure, cycle ergometer test to evaluate cardiovascular fitness, an echocardiography to determine epicardial fat thickness, a dual energy x-ray absorptiometry (DEXA) scan to assess body fat, lean mass and bone density, indirect calorimetry for resting metabolic rate, physical activity profile and total energy expenditure determined by Sense Wear Armband (SWA) accelerometer (7days), food consumption estimate with 3 days dairy, questionnaires addressing sociodemographic and psychosocial characteristics, diabetes self-care (SDCA questionnaire), a blood and urine collection for diabetes control, hepatic steatosis biochemical score, detailed lipids, hormonal and inflammatory profile and finally microalbuminuria. The body composition will also be measured by impedancemetry and BOD-POD.

Participants will then be randomly assigned to one of the three groups of the study :

Group 1: Counseling for physical activity and healthy eating Group 2: Structured diet intervention (caloric restriction) and counseling for physical activity Group 3: Structured diet intervention (caloric restriction) and structured exercise training program (aerobic and resistance training).

Group 1: participants will attend one visit with the dietician (30mn) and the physical activity specialist (30mn) when they will be given Canadian guidelines pamphlets for physical activity and food consumption. They will also receive a phone call once a month to discuss about issues in guidelines following.

Group 2: participants will attend one visit with the physical activity specialist (30mn) when they will receive the physical activity guidelines. Monthly phone call will be make to discuss about issues in physical activity guidelines following. These individuals will also be enrolled in a supervised caloric restriction program. They will have to visit the dietician once a week for the first months and then twice a month for 3 months. The diet intervention will focus on a low fat diet. At each session participants will be weighed and taken the blood pressure.

Group 3: participants will attend diet intervention as described for group 2. They will also follow a supervised exercise program three days per week for 4 months. The exercise training is an interval high intensity aerobic (85-90% Heart rate reserve) program with resistance exercises (15RM, 2-3 repetitions). Each session will last one hour. At the end of month 1, 2, and 3, all participants will receive the SWA armband for 7 days to record physical activity and estimate energy expenditure.

At the end of Month 4, all participants will attend a study visit for repeat baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 27-40 kg/m2
* Type 2 diabetes diagnosed since at least 3 months
* High risk of cardiovascular disease : Framingham global cardiovascular risk score for 10 years > 15% or 2 or more of the following risk factors: age > 50years, dyslipidemia or treatment, high blood pressure or treatment, pathologic microalbuminuria or established proteinuria, currently smoking, family history of early cardiovascular disease (< 60 years), inactivity or high waist circumference according to IDF criteria
* HbA1c : 6.0-10.0%
* Stable weight for last 3 months (±3kg) reported or documented
* Stable treatment for diabetes. 4 weeks: blood pressure and dyslipidemia medications. 3 months: glitazones and weight loss drugs the treatment that will be maintained at the same dose during the study; insulin will have been introduced since 4 months at least and previous month dose should be stable defined as a 10% variation or less of total daily units.

Exclusion Criteria:

* Pregnancy, breastfeeding
* Type 1 diabetes
* Secondary diabetes (e.g cystic fibrosis, steroid induced, etc.)
* Recurrent, hypoglycemia without precursor signs or severe hypoglycemia occurred ≥ 2 times for last 12 months
* Renal failure , creatinine clearance < 40 ml/min (MDRD)
* Severe retinopathy or neuropathy that can contra-indicate exercise or expose patient to high risk of complications (e.g wound)
* NYHA classification class III or IV of cardiac insufficiency
* Established coronaropathy
* Non stable ventricular or supra-ventricular arrythmia
* Severe limb atherosclerosis or previous amputation
* Recent (< 12 months) diagnosis of cancer excepted thyroid and skin
* Major mental disease
* Drugs with established effects on weigh such as megace®

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Total fat mass | month 4
  Total fat mass (kg) assessed by Dual X-Ray absoptiometry (DXA)

SECONDARY OUTCOMES:
Diabetes control | month 4
  A1c and fasting plasma glucose
Epicardial fat | month 4
  Epicardial fat thickness measured by simplified cardiac echography
Body composition | month 4
  Body composition : trunkal fat mass, apendicular fat mass, lean body mass and estimated visceral fat mass determined by DXA
Energy consumption | month 4
  Energy consumption : as measured by total calories consumed using a three non consecutive days food journal. The three days should include one week-end day.
Resting metabolic rate | month 4
  Resting metabolic rate determined by indirect calorimetry.
Total energy expenditure | month 2,3,4
  Total energy expenditure estimated from 7 days accelerometer data (Senwear Armband accelerometer).
Physical activity energy expenditure | month 2,3,4
  Physical activity energy expenditure estimated from 7 days accelerometer data (Senwear Armband accelerometer).
Muscle strength | month 4
  upper and lower body strength using 1-RM technique
Cardiorespiratory fitness | month 4
  Participants will perform a graded exercise test on a cycle ergometer to voluntary exhaustion. Peak oxygen consumption (VO2peak) will be considered to be the highest value obtained during the test.
Lipid profile | month 4
  Total cholesterol, LDL-Cholesterol, HDL-cholesterol (HDL-C), Triglycerides, Apolipoprotein B, ratios TG/HDL-C and Total cholesterol/HDL-C will be determined with fasting veinous blood sample
Biochemical hepatic steatosis score | month 4
Blood pressure | month 4
  systolic and diastolic blood pressure
Hormonal profile | month 4
Inflammatory profile | month 4
Psychosocial profile | month 4
  questionnaire addressing : body esteem, self-esteem, stress, dietary restraint, disinhibition, hunger, quality of life, self-efficacy,perceived benefits, perceived risks
Diabetes self-care | month 4
  Summary of diabetes care activities (SDCA) questionnaire
visceral fat thickness | month 4

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de Recherches Cliniques de Montreal; Antony Karelis, PhD, Study Chair — Université de Québec à Montréal; Denis Prud'Homme, MD, Msc, Study Chair — University of Ottawa; Eric Doucet, PhD, Study Chair — University of Ottawa
Locations (1):
- Institut de recherches cliniques de Montréal (IRCM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Leroux-Stewart J, Elisha B, Tagougui S, Suppere C, Bernard S, Mircescu H, Desjardin K, Messier V, Iacobellis G, Rabasa-Lhoret R. Effect of caloric restriction with or without physical activity on body composition and epicardial fat in type 2 diabetic patients: A pilot randomized controlled trial. Nutr Metab Cardiovasc Dis. 2021 Mar 10;31(3):921-929. doi: 10.1016/j.numecd.2020.11.005. Epub 2020 Nov 13. PMID 33549453